CLINICAL TRIAL: NCT02580916
Title: Use of the Skin Cancer Quality of Life Impact Tool (SCQOLIT) - a Feasibility Study in Non-melanoma Skin Cancer
Brief Title: Utility of the Skin Cancer Quality of Life Impact Tool
Acronym: SCQOLIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Rubeta Matin, Consultant Dermatologist, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11054
Record Dates: First submitted 2015-08-25; First posted 2015-10-20 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Skin Neoplasm; Squamous Cell Carcinoma; Basal Cell Carcinoma
Keywords: non-melanoma skin cancer; outcome assessment; quality of life
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Squamous Cell; Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Postal) (Experimental): These are patients who will be identified from the histological diagnosis of their skin cancer by members of the direct care team and deemed 'low risk'; SCQOLIT questionnaires will be administered by post.
  Interventions: Other: SCQOLIT questionnaire
- Group 2 (Clinic-based) (Experimental): These are patients who will be identified from the histological diagnosis of their skin cancer by members of the direct care team, for whom all aspects of the study will be conducted in the Dermatology clinic. SCQOLIT questionnaires will be administered according to the protocol.
  Interventions: Other: SCQOLIT questionnaire
- Group 3 (Interviews) (No Intervention): A Qualitative Researcher (Co-Investigator) will undertake structured interviews with approximately 20 patients from both Group 1 and 2. Potential participants will be invited to volunteer their contact details at the time of consent to the Questionnaire study. This is optional; they may refuse to do so and still take part in the main questionnaire study. The patient will then be contacted by the Qualitative Researcher (Co-Investigator) at a later date and subsequently consented for the interview.
- Group 4 (Clinician focus group) (No Intervention): We aim to discuss the project at the end of the study period in the same setting, to establish staff perspectives on the study, to establish usefulness of the SCQOLIT tool and to identify any barriers to implementation.

INTERVENTIONS:
Other: SCQOLIT questionnaire — Participants will be invited to complete the SCQOLIT and EQ-5D (used for comparison purposes, given its widespread use in other healthcare contexts in the UK) questionnaires [Appendices C & D) at:
  1. baseline (after histological diagnosis of a NMSC is confirmed - both Groups)
  2. 3 months - either by postal (Group 1) or face-to-face (Group 2) dependent on whether the patient is returning to the Dermatology clinic for routine follow-up
  3. at 6-9 months in the dermatology clinic if the patient is deemed high risk (squamous cell carcinoma with high risk clinicopathological features as listed by the National British Association Dermatologists Multiprofessional Guidelines for management of SCC) (Group 2 only)
  Arms: Group 1 (Postal); Group 2 (Clinic-based)

SUMMARY:
Background:

Patient-reported outcome measures (PROMs) provide validated evidence of health and quality of life (QoL) from the patient perspective. Several national PROMs programmes have been implemented in the National Health Service - specifically for common elective procedures. Local implementation is varied across settings and populations. The incidence of non-melanoma skin cancer (NMSC) is rapidly increasing, posing considerable burden on UK healthcare resources, yet there is limited evidence of use of PROMs in NMSC and little information about patients' perceived health and QoL.

Objectives:

This study will explore feasibility of implementing a skin cancer-specific PROM - Skin Cancer Quality of Life Impact Tool (SCQOLIT) for NMSC.

Methods:

Three hundred patients with a pathological diagnosis of NMSC undergoing all treatment modalities will be recruited to complete SCQOLIT questionnaires at baseline, at 3, 6 and 9 months. Participation and response rates, missing data and individual change scores will be analysed. Staff and patients will be interviewed to explore acceptability and feasibility of collecting PROMs data.

Results:

Interim results of the project to date will be presented. Feasibility will be assessed by evaluating number of eligible patients, number of consenting patients, reasons for not consenting and participant number. Individual longitudinal change in scores, response rates and psychometric properties of the SCQOLIT will be reported.

Implications:

Acceptability and feasibility of the SCQOLIT tool has never been rigorously assessed in Dermatology clinics. A validated NMSC-specific PROM would help standardize multi-centred trials, allow robust evaluation of quality of care and more appropriately direct healthcare resources to improve QoL in patients with NMSC.

DETAILED DESCRIPTION:
Background:

Skin cancer is the most rapidly increasing cancer type in fair-skinned populations worldwide. Although non-melanoma skin cancer (NMSC) are rarely life threatening, both disease and treatments can be associated with substantial morbidity and confer significant financial burden to the National Health Service (NHS). Consequently, the British Association of Dermatologists (BAD) commissioned the Patient-reported Outcomes Measurement Group, Oxford to review the evidence for PROMs for skin cancer. The authors concluded that cancer-specific quality of life (QOL) questionnaires appeared more sensitive than generic PROMs e.g. the Dermatology Life Quality Index (DLQI), in capturing relevant QOL issues. In the NMSC population, these issues include scarring, disfigurement, anxiety and fear of future skin cancers.

One skin cancer-specific PROM that was evaluated was the Skin Cancer Quality of Life Impact Tool (SCQOLIT). The SCQOLIT is a ten-item instrument developed specifically for patients with non-metastatic skin cancer, which has demonstrated evidence in favour of reproducibility, validity, internal consistency but requires further evaluation.

The decision to evaluate the SCQOLIT in this study, includes its similarity in overall format and brevity to that of the DLQI which is a PROM now widely used in routine medical dermatology clinical practice. The SCQOLIT takes less than five minutes for the patient to complete and has a similar score calculation to the DLQI. Acceptability and feasibility of this tool has never been rigorously assessed in Dermatology clinics. Studies evaluating PROMs in NMSC have been largely assessed in relation to surgical treatments yet basal cell carcinoma can be effectively treated using medical treatments e.g. topical immunomodulators and photodynamic therapy, and to date, PROMs have not been investigated in these sub-populations.

Justification:

This feasibility study is designed to evaluate the SCQOLIT questionnaire, and aims to establish its utility and impact in patients with NMSC. The investigators will assess both patient and clinician acceptability of the SCQOLIT questionnaire tool and hope to identify any unmet needs, which can potentially inform future clinical decisions and/or service planning.

Study design:

Participants:

All patients referred to Dermatology Tumour outpatient clinics with a clinically suspected NMSC.

There will be four categories of participants, Groups 1 - 3 are participants with a new diagnosis of NMSC (primary or recurrent) on any site of the body:

Group 1 (Postal) - this will include those patients with a 'low risk' NMSC (namely basal cell carcinoma)

Group 2 (Clinic-based) - this will include those patients with a 'moderate to high risk' NMSC (namely SCC or other rare NMSC)

Group 3 (Interview) - these will be volunteers selected from Groups 1 and 2.

Group 4 (Focus Group: Clinicians) - this will include any Dermatology staff member who is involved in consenting and collecting PROMS data and has a role for direct care of patients attending Dermatology outpatient clinics.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 yrs old
* All patients with a histopathological diagnosis of NMSC (primary or recurrent disease)
* All treatments used for NMSC will be included; excision, shave excision, curettage and cautery, Mohs micrographic surgery, photodynamic therapy and topical treatments e.g. imiquimod cream.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Concurrent internal malignancy as this is likely to significantly influence QOL.
* Patients referred onwards to other specialties for management of their skin cancer e.g. Plastic surgeons / Clinical oncology.
* Other significant dermatological diseases e.g. severe inflammatory or blistering skin conditions as this may influence QOL.
* Inability to consent for themselves.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2015-07; Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
SCQOLIT questionnaire response rates | 2 years
  Quantitative analysis of patient participation rates in the study, questionnaire response rates and number of missing values.
Qualitative analysis of patient and staff preferences, views and experiences | 2 years
  Analysis of structured interviews and focus group to establish acceptability of SCQOLIT tool

SECONDARY OUTCOMES:
Construct validity of SCQOLIT tool | 2 years
  Measure of psychometric property of SCQOLIT
Responsiveness of SCQOLIT tool | 2 years
  Measure of psychometric property of SCQOLIT
Differences in scores from baseline to follow-up | 2 years
  Measure of psychometric property of SCQOLIT - clinically important difference. A statistical analysis of the differences in scores will be calculated.
Proportion of responses at the uppermost and lowermost end of the scale | 2 years
  Measure of psychometric property of SCQOLIT - floor and ceiling effect - to evaluate the range of scores and to determine how many responses are at the highest and lowest scores.
Intra- and inter- participant change in scores | 2 years
  Measure of psychometric property of SCQOLIT

CONTACTS AND LOCATIONS:
Overall Officials: Rubeta N Matin, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Churchill Hospital, Headington, Oxford, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT02580916/Prot_SAP_000.pdf